CLINICAL TRIAL: NCT03351205
Title: Randomized, Controlled Trial to Assess the Efficacy of Estrogen Therapy Combined With Disposable Balloon Uterine Stent and Dried Biological Amnion Graft in the Prevention of Adhesion Reformation After Hysteroscopic Adhesiolysis
Brief Title: The Efficacy of Estrogen Therapy Against Adhesion Reformation After Hysteroscopic Adhesiolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: No.6-20171120
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Intrauterine Adhesion
Keywords: Asherman syndrome; hysteroscopy; uterine stent; Estrogen; Amnion; Hysteroscopic Adhesiolysis
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uterine cavity barrier only (Experimental): patients, who are with IUA, treated by uterine application of disposable balloon uterine stent + amnion membrane following hysteroscopic adhesiolysis.
  Interventions: Device: disposable balloon uterine stent; Procedure: dried biological amnion graft
- hormone (Experimental): patients, who are with IUA, treated by uterine application of disposable balloon uterine stent+ amnion membrane+hormones (estradiol valerate tablets+dydrogesterone Tablets) following hysteroscopic adhesiolysis.
  Interventions: Device: disposable balloon uterine stent; Procedure: dried biological amnion graft; Drug: estradiol valerate tablets+dydrogesterone tablets

INTERVENTIONS:
Device: disposable balloon uterine stent — The disposable balloon uterine stent is heart-shaped that resembled the shape of the uterine cavity and could fully separate the two sides of the uterine wall and the corners of the uterus compare to Foley catheter.
Procedure: dried biological amnion graft — Uterine application of dried biological amnion graft following hysteroscopic adhesiolysis.
  Other Name: Human amnion membrane
  Other Names: amnion membrane
Drug: estradiol valerate tablets+dydrogesterone tablets — oral estradiol valerate tablets+dydrogesterone tablets
  Other Names: Progynova+dydrogesterone
  Arms: hormone

SUMMARY:
Asherman's syndrome is characterized by the presence of intrauterine adhesions (IUA) as well as symptoms such as amenorrhea, hypomenorrhea, pelvic pain, and infertility. The gold standard for the treatment of intrauterine adhesions is hysteroscopic intrauterine adhesions. The recurrence of intrauterine adhesions is a major challenge in clinical practice. Intrauterine balloon has been used for the prevention of intrauterine adhesions. It has been reported that dried biological amnion graft was used to prevent adhesion after the operation of intrauterine adhesions. Estrogen is also used for postoperative prevention of intrauterine adhesions. Intrauterine balloon can reduce the recurrence of adhesions after operation. Disposable balloon uterine stent，which is an innovative intrauterine balloon，is specially designed to fit into the cavity of the uterus. Does Disposable balloon uterine stent and amniotic products combine estrogen therapy improve clinical outcomes? Therefore, this study was conducted.

DETAILED DESCRIPTION:
Allocation: Randomized Endpoint Classification: Efficacy Study Intervention Model: Parallel Assignment Masking: Double (participant and outcomes Assessor) Primary Purpose: Prevention

ELIGIBILITY:
Inclusion Criteria:

* age 20-40 years；
* previously diagnostic hysteroscopy confirmed adhesion score >5， according to the American Fertility Society （AFS）classification of IUA；
* complains of menstruation disorder and reproductive dysfunction；
* informed consent.

Exclusion Criteria:

* premature menopause,
* presence of other intrauterine lesions (e.g. polyps, myoma, septa), and
* presence of severe intercurrent illness (e.g. systemic disease, coagulative disorders, severe kidney and liver diseases),
* adhesions limited to the lower uterine cavity or the cervical canal.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-21 (Estimated); Primary Completion 2018-11-21 (Estimated); Study Completion 2018-11-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of adhesion information | Within the first 3 months after surgery
  Intrauterine adhesions under hysteroscopy

SECONDARY OUTCOMES:
Menstruation Pattern | Within the first 3 months after surgery
  menstrual volume which was assessed by pictorial blood loss assessment chart
The change of AFS score | Within the first 3 months after surgery
  he American Fertility Society ( AFS ) scoring system (1988 version). Scores of 1-4, 5-8, and 9-12 were mild, moderate, and severe adhesions, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Duan Hua, MD, Study Chair — Beijing Obstetrics and Gynecology Hospital
Locations (1):
- Beijing Obstetrics and Gynecology Hospital，Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes